## Incentives for Postnatal Care Demand NCT02936869

July 7, 2016

## **Proposed Empirical Models**

## 1. Average effect of incentives on early PNC referrals

I identify the intention-to-treat effect of incentives on the proportion of TBA deliveries referred for postnatal care within 48 hours of delivery (early PNC).

$$y_{ii} = \beta_0 + \beta_1 * T + X_{ii} + \varepsilon_{ii}$$

Where:

- $y_{ij}$  is proportion of delivery clients or neonates (all, with or without delivery complications) referred by TBA i, in village j for early PNC;
- T is a dummy variable indicating if the TBA is in the treatment arm;
- $X_{ij}$  is a set of baseline TBA covariates;
- $\beta_1$  is the coefficient of interest and gives the average mean difference in proportion of TBA clients referred between the treatment and the control arm.

## 2. Heterogeneity in the effect of incentives on early PNC referrals

I also identify interactions between incentives and baseline TBA characteristics (considered proxies for social preferences) in order to clarify pathways through which the intervention might have worked. I specify a series of equations:

$$y_{ij} = \beta_0 + \beta_1 * T + \beta_2 * T * V ar_{ij} + V ar_{ij} + X_{ij} + \varepsilon_{ij}$$

Where:

- $Var_{ij}$  is a binary baseline characteristic for TBA i in village j previously included in  $X_{ij}$ ;
- $\beta_1$  is interpreted as the treatment effect when  $Var_{ij} = 0$ ;
- $\beta_2$  is the additional effect of  $Var_{ii}$